CLINICAL TRIAL: NCT03042234
Title: Effects of High-intensity Interval Training on Cardiorespiratory Performance and Substrate Oxidation in Insulin-resistant and Insulin-sensitive Obese Adolescents: A Before-and-after Clinical Study
Brief Title: HIT in Insulin-resistant and Insulin-sensitive Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, JULIANA MONIQUE LINO, Principal investigator Juliana Monique Lino Aparecido, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: japarecido; 34634414.5.0000.5479 (Registry Identifier: CAAE); 1.227.250 (Other: Number of opinion)
Record Dates: First submitted 2017-01-30; First posted 2017-02-03 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Insulin-resistant; Adolescents
Keywords: Obesity; Insulin-resistant; Adolescents; High-intensity interval training
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Insulin-resistant (Experimental): Insulin-resistant obese adolescents
  Interventions: Other: Group Insulin-Resistant; Other: Group Insulin-Sensitive
- Group Insulin-sensitive (Experimental): Insulin-sensitive obese adolescents
  Interventions: Other: Group Insulin-Resistant; Other: Group Insulin-Sensitive

INTERVENTIONS:
Other: Group Insulin-Resistant — High intensity interval training: 3 to 6 sets of 60-second sprints at 100% of the peak velocity interspersed by a 3-min active recovery period.
  Other Names: Insulin-resistant obese adolescents
Other: Group Insulin-Sensitive — High intensity interval training: 3 to 6 sets of 60-second sprints at 100% of the peak velocity interspersed by a 3-min active recovery period.
  Other Names: Insulin-sensitive obese adolescents

SUMMARY:
Evaluate the effects of HIT on the cardiorespiratory performance and substrate oxidation of insulin-resistant and insulin-sensitive obese adolescents.

DETAILED DESCRIPTION:
Objective: To evaluate the effect of high-intensity interval training (HIT) on the cardiorespiratory performance and substrate oxidation pattern in insulin-resistant and insulin-sensitive obese adolescents.

ELIGIBILITY:
Criteria

Inclusion Criteria:

* aged 12-16 years
* with a body mass index z-score (zBMI) ≥ + 2SD
* puberty stage > 3
* the boys and girls had to present a minimum physical fitness, according to the International Physical Activity Questionnaire (IPAQ), according to the activity performed during the last week and confirmed this using the peak cardiopulmonary test (VO2).

Exclusion Criteria:

* individuals undergoing drug treatment for weight control;
* indiviudals who had cardiac, orthopedic, respiratory or renal problems, diabetes, uncontrolled hypertension, genetic syndrome or hormonal abnormalities.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2017-07-08 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
rate of Peak oxygen consumption (VOpeak) | 4 weeks
  The cardiopulmonary test protocol for determination the VOpeak (ml/kg/min) included running on a treadmill (Model ATL, Inbrasport Ltda; Brazil) at a speed of 4 km/h with 1 km/h increments every minute until the participant showed exhaustion.
  We evaluated ventilatory parameters on a gas analyzer (model VO2000; Inbrasport Ltda; Brazil).
rate of Intensity at first ventilatory anaerobic threshold (VAT1) | 4 weeks
  The cardiopulmonary test protocol included running on a treadmill (Model ATL, Inbrasport Ltda; Brazil) at a speed of 4 km/h with 1 km/h increments every minute until the participant showed exhaustion.
  We evaluated ventilatory parameters on a gas analyzer (model VO2000; Inbrasport Ltda; Brazil).We determined VAT1 (ml/kg/min) using the V-slope method of Beaver et al.
rate of Peak Heart rate | 4 weeks
  The cardiopulmonary test protocol included treadmill running (Model ATL, Inbrasport Ltda; Brazil). speed of 4 km / h with increments of 1 km / h every minute until the participant shows exhaustion.
rate of carbohydrate oxidation | 4 weeks
  The substrate oxidation pattern protocol included treadmill running (Model ATL, Inbrasport Ltda; Brazil),during continuous exercise of submaximal intensity (45 minutes of treadmill running at the intensity of the first ventilatory anaerobic threshold).
rate of lipid oxidation | 4 weeks
  The substrate oxidation pattern protocol included treadmill running (Model ATL, Inbrasport Ltda; Brazil),during continuous exercise of submaximal intensity (45 minutes of treadmill running at the intensity of the first ventilatory anaerobic threshold).

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Monique Lino Aparecido, Principal Investigator — Faculdade de Ciências Médicas da Santa Casa de São Paulo
Locations (3):
- Brazil (3):
  - Santa Casa of Sao Paulo School, São Paulo
  - Emef Angelina Maffei Vita, São Paulo
  - Emef Plinio Queroz, São Paulo

REFERENCES:
- [Background] ROSSETTI, MB; BRITO, RR; NORTON, RC. Prevenção primária de doenças cardiovasculares na obesidade infatojuvenil: efeito anti-inflamatório do exercício físico. Rev Bras Med Esporte. 2009
- [Background] Corte de Araujo AC, Roschel H, Picanco AR, do Prado DM, Villares SM, de Sa Pinto AL, Gualano B. Similar health benefits of endurance and high-intensity interval training in obese children. PLoS One. 2012;7(8):e42747. doi: 10.1371/journal.pone.0042747. Epub 2012 Aug 6. PMID 22880097
- [Background] KLOSTER, R & LIBERALI, R. Emagrecimento: composição da dieta e exercício físico. Rev Bras Nutr Esportiva. 2012 set-out; 11(2):288-306
- [Background] FOUREAUX, G; PINTO, KMC; DÂMASO, A. Efeito do consumo excessivo de oxigênio após exercício e da taxa metabólica de repouso no gasto energético. Rev Bras Med Esporte. 2006 nov-dez; 12(6):393-398.
- [Background] AMERICAN COLLEGE OF SPORTS MEDICINE - ACSM. ACSM's Guidelines for Exercise Testing and Prescription. 8ª edição. Baltimore: Williams & Wilkins, 2009.
- [Background] Aucouturier J, Rance M, Meyer M, Isacco L, Thivel D, Fellmann N, Duclos M, Duche P. Determination of the maximal fat oxidation point in obese children and adolescents: validity of methods to assess maximal aerobic power. Eur J Appl Physiol. 2009 Jan;105(2):325-31. doi: 10.1007/s00421-008-0907-3. Epub 2008 Nov 12. PMID 19002708
- [Background] MARQUEZI, ML. Adaptações decorrentes do exercício cardiorrespiratório sobre a oxidação de lipídeos: exercício aeróbio. Rev Mackenzie de Educação Física e Esporte. 2010; 9(1):32-35.
- [Background] Achten J, Gleeson M, Jeukendrup AE. Determination of the exercise intensity that elicits maximal fat oxidation. Med Sci Sports Exerc. 2002 Jan;34(1):92-7. doi: 10.1097/00005768-200201000-00015. PMID 11782653
- [Background] Achten J, Jeukendrup AE. Relation between plasma lactate concentration and fat oxidation rates over a wide range of exercise intensities. Int J Sports Med. 2004 Jan;25(1):32-7. doi: 10.1055/s-2003-45231. PMID 14750010
- [Background] MARQUEZI, ML; DUARTE, L; SCHWARTZ, J; SOUSA, PCR. Variabilidade interindividual da oxidação de substratos durante o exercício. Rev Mackenzie de Educação Física e Esporte. 2009; 8(1): 3-19.
- [Background] Carey DG. Quantifying differences in the "fat burning" zone and the aerobic zone: implications for training. J Strength Cond Res. 2009 Oct;23(7):2090-5. doi: 10.1519/JSC.0b013e3181bac5c5. PMID 19855335
- [Background] Braun B, Sharoff C, Chipkin SR, Beaudoin F. Effects of insulin resistance on substrate utilization during exercise in overweight women. J Appl Physiol (1985). 2004 Sep;97(3):991-7. doi: 10.1152/japplphysiol.00231.2004. Epub 2004 May 7. PMID 15133003
- [Background] Blaak EE, van Aggel-Leijssen DP, Wagenmakers AJ, Saris WH, van Baak MA. Impaired oxidation of plasma-derived fatty acids in type 2 diabetic subjects during moderate-intensity exercise. Diabetes. 2000 Dec;49(12):2102-7. doi: 10.2337/diabetes.49.12.2102. PMID 11118013
- [Background] Borghouts LB, Wagenmakers AJ, Goyens PL, Keizer HA. Substrate utilization in non-obese Type II diabetic patients at rest and during exercise. Clin Sci (Lond). 2002 Dec;103(6):559-66. doi: 10.1042/cs1030559. PMID 12444908
- [Background] Perez-Martin A, Dumortier M, Raynaud E, Brun JF, Fedou C, Bringer J, Mercier J. Balance of substrate oxidation during submaximal exercise in lean and obese people. Diabetes Metab. 2001 Sep;27(4 Pt 1):466-74. PMID 11547220
- [Background] Gibala MJ, Little JP, Macdonald MJ, Hawley JA. Physiological adaptations to low-volume, high-intensity interval training in health and disease. J Physiol. 2012 Mar 1;590(5):1077-84. doi: 10.1113/jphysiol.2011.224725. Epub 2012 Jan 30. PMID 22289907
- [Background] Donnelly JE, Blair SN, Jakicic JM, Manore MM, Rankin JW, Smith BK; American College of Sports Medicine. American College of Sports Medicine Position Stand. Appropriate physical activity intervention strategies for weight loss and prevention of weight regain for adults. Med Sci Sports Exerc. 2009 Feb;41(2):459-71. doi: 10.1249/MSS.0b013e3181949333. PMID 19127177
- [Background] Burgomaster KA, Howarth KR, Phillips SM, Rakobowchuk M, Macdonald MJ, McGee SL, Gibala MJ. Similar metabolic adaptations during exercise after low volume sprint interval and traditional endurance training in humans. J Physiol. 2008 Jan 1;586(1):151-60. doi: 10.1113/jphysiol.2007.142109. Epub 2007 Nov 8. PMID 17991697
- [Background] Talanian JL, Holloway GP, Snook LA, Heigenhauser GJ, Bonen A, Spriet LL. Exercise training increases sarcolemmal and mitochondrial fatty acid transport proteins in human skeletal muscle. Am J Physiol Endocrinol Metab. 2010 Aug;299(2):E180-8. doi: 10.1152/ajpendo.00073.2010. Epub 2010 May 18. PMID 20484014
- [Background] Tjonna AE, Lee SJ, Rognmo O, Stolen TO, Bye A, Haram PM, Loennechen JP, Al-Share QY, Skogvoll E, Slordahl SA, Kemi OJ, Najjar SM, Wisloff U. Aerobic interval training versus continuous moderate exercise as a treatment for the metabolic syndrome: a pilot study. Circulation. 2008 Jul 22;118(4):346-54. doi: 10.1161/CIRCULATIONAHA.108.772822. Epub 2008 Jul 7. PMID 18606913
- [Background] Talanian JL, Galloway SD, Heigenhauser GJ, Bonen A, Spriet LL. Two weeks of high-intensity aerobic interval training increases the capacity for fat oxidation during exercise in women. J Appl Physiol (1985). 2007 Apr;102(4):1439-47. doi: 10.1152/japplphysiol.01098.2006. Epub 2006 Dec 14. PMID 17170203
- [Background] Perry CG, Heigenhauser GJ, Bonen A, Spriet LL. High-intensity aerobic interval training increases fat and carbohydrate metabolic capacities in human skeletal muscle. Appl Physiol Nutr Metab. 2008 Dec;33(6):1112-23. doi: 10.1139/H08-097. PMID 19088769
- [Background] Little JP, Safdar A, Wilkin GP, Tarnopolsky MA, Gibala MJ. A practical model of low-volume high-intensity interval training induces mitochondrial biogenesis in human skeletal muscle: potential mechanisms. J Physiol. 2010 Mar 15;588(Pt 6):1011-22. doi: 10.1113/jphysiol.2009.181743. Epub 2010 Jan 25. PMID 20100740
- [Background] Little JP, Safdar A, Bishop D, Tarnopolsky MA, Gibala MJ. An acute bout of high-intensity interval training increases the nuclear abundance of PGC-1alpha and activates mitochondrial biogenesis in human skeletal muscle. Am J Physiol Regul Integr Comp Physiol. 2011 Jun;300(6):R1303-10. doi: 10.1152/ajpregu.00538.2010. Epub 2011 Mar 30. PMID 21451146
- [Background] Baquet G, Gamelin FX, Mucci P, Thevenet D, Van Praagh E, Berthoin S. Continuous vs. interval aerobic training in 8- to 11-year-old children. J Strength Cond Res. 2010 May;24(5):1381-8. doi: 10.1519/JSC.0b013e3181d1575a. PMID 20440122
- [Background] de Onis M, Onyango AW, Borghi E, Siyam A, Nishida C, Siekmann J. Development of a WHO growth reference for school-aged children and adolescents. Bull World Health Organ. 2007 Sep;85(9):660-7. doi: 10.2471/blt.07.043497. PMID 18026621
- [Background] TANNER JM. Growth at adolescence. Oxford: Blackwell Scientific Pub; 1962.
- [Background] MATSUDO, SM; ARAÚJO, TL; MATSUDO, VKR; ANDRADE, DR; ANDRADE, EL; OLIVEIRA, LC; et al. Questionário Internacional de Atividade Física (IPAQ): estudo de validade e reprodutibilidade no Brasil. Rev Bras Ativ Saude. 2001;10:5-18.
- [Background] Pereira CA, Sato T, Rodrigues SC. New reference values for forced spirometry in white adults in Brazil. J Bras Pneumol. 2007 Jul-Aug;33(4):397-406. doi: 10.1590/s1806-37132007000400008. English, Portuguese. PMID 17982531
- [Background] Caiozzo VJ, Davis JA, Ellis JF, Azus JL, Vandagriff R, Prietto CA, McMaster WC. A comparison of gas exchange indices used to detect the anaerobic threshold. J Appl Physiol Respir Environ Exerc Physiol. 1982 Nov;53(5):1184-9. doi: 10.1152/jappl.1982.53.5.1184. PMID 7174412
- [Background] WASSERMAN K, MCILROY MB. DETECTING THE THRESHOLD OF ANAEROBIC METABOLISM IN CARDIAC PATIENTS DURING EXERCISE. Am J Cardiol. 1964 Dec;14:844-52. doi: 10.1016/0002-9149(64)90012-8. No abstract available. PMID 14232808
- [Background] Bhambhani Y, Singh M. Ventilatory thresholds during a graded exercise test. Respiration. 1985;47(2):120-8. doi: 10.1159/000194758. PMID 4001567
- [Background] Gmada N, Marzouki H, Haboubi M, Tabka Z, Shephard RJ, Bouhlel E. Crossover and maximal fat-oxidation points in sedentary healthy subjects: methodological issues. Diabetes Metab. 2012 Feb;38(1):40-5. doi: 10.1016/j.diabet.2011.07.004. Epub 2011 Sep 25. PMID 21944864
- [Background] Cheneviere X, Malatesta D, Peters EM, Borrani F. A mathematical model to describe fat oxidation kinetics during graded exercise. Med Sci Sports Exerc. 2009 Aug;41(8):1615-25. doi: 10.1249/MSS.0b013e31819e2f91. PMID 19568198
- [Background] Lanzi S, Codecasa F, Cornacchia M, Maestrini S, Salvadori A, Brunani A, Malatesta D. Fat oxidation, hormonal and plasma metabolite kinetics during a submaximal incremental test in lean and obese adults. PLoS One. 2014 Feb 11;9(2):e88707. doi: 10.1371/journal.pone.0088707. eCollection 2014. PMID 24523934